CLINICAL TRIAL: NCT07296068
Title: Can Acute Photobiomodulation Improve Balance and Cognition in Individuals With Ataxia: a Pilot Feasibility Placebo Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMB Ataxia pilot feasibility s
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ataxia
MeSH Terms: conditions — Ataxia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Comparator: Sham photobiomodulation (Placebo Comparator): Sham photobiomodulation. The sham device will follow the same protocol but without active light emission.
  Interventions: Other: Sham photobiomodulation
- Photobiomodulation (Experimental): Acute photobiomodulation Twenty-four-minute photobiomodulation stimulation (twelve minutes at 670 nm followed by twelve minutes at 810 nm).
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Photobiomodulation
  Arms: Photobiomodulation
Other: Sham photobiomodulation — The sham device will follow the same protocol but without active light emission.
  Arms: Sham Comparator: Sham photobiomodulation

SUMMARY:
Cerebellar ataxias cause progressive impairments in balance, gait coordination, motor timing, and cognitive functions such as attention and executive control (Buckner, 2013; Salmi et al., 2010; Timmann & Daum, 2007). These symptoms substantially reduce independence and quality of life, and current treatments remain limited. There is an urgent need for safe, low-burden interventions that can support everyday functioning and potentially enhance compensatory neural processes.

Transcranial photobiomodulation (tPBM) uses red and near-infrared light (600-1100 nm) to modulate mitochondrial cytochrome-c oxidase, increasing ATP production, reducing oxidative stress, and improving cerebral blood flow (Hamblin, 2016; Salehpour et al., 2019). Several studies show that tPBM can acutely improve cognitive performance and motor control in both healthy adults and clinical groups (Barrett & Gonzalez-Lima, 2013; Chan et al., 2019; Henderson & Morries, 2017). A growing neurobiological literature suggests that light can penetrate posterior cortical areas sufficiently to modulate networks involving cerebellar-cortical loops (Jagdeo et al., 2012).

Importantly for ataxia, preliminary work shows that tPBM may acutely improve balance stability and gait metrics in older adults and patients with neurological conditions (Moro et al., 2022; Shin et al., 2021). In our own laboratory, we have observed immediate improvements in sway range and cognitive control in older adults after a 24-minute tPBM session applied over midline and posterior scalp regions. These medium to large size effects are consistent with enhanced sensorimotor integration and improved control of attention in distracting environments.

Given that individuals with cerebellar ataxia experience both motor incoordination and difficulties in maintaining cognitive stability under distracting conditions, tPBM is a promising non-pharmacological intervention worth preliminary investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years (inclusive)
* Diagnosis of ataxia
* Able to walk independently for at least 5 minutes, with or without an assistive device
* Able to stand safely for balance testing, with or without an assistive device
* Hemodynamically stable (stable blood pressure and heart rate at rest)
* On a stable medication regimen for ≥4 weeks prior to enrolment
* Sufficient vision and hearing (with usual aids if required) to complete balance and cognitive assessments
* Able to complete study questionnaires and cognitive tasks (with assistance for reading/writing if required)
* Able and willing to provide written informed consent

Exclusion Criteria:

* Current or past history of head injury
* Use of medications acting on the central nervous system
* Active skin conditions on the forehead or scalp
* Any other major neurological disorder that could independently affect balance or cognition
* Ongoing brain stimulation therapy
* History of migraines
* Sensitive skin, allergies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
n-1-back (deviation) | Baseline
  The n-1-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-1 trials earlier.
n-1-back (deviation) | 1 hour
  The n-1-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-1 trials earlier.

SECONDARY OUTCOMES:
n-2-back (deviation) | Baseline
  The n-2-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-2 trials earlier.
n-2-back (deviation) | 1 hour
  The n-2-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-2 trials earlier.
n-1-back (post-deviation) | Baseline
  The n-1-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-1 trials earlier.
n-1-back (post-deviation) | 1 hour
  The n-1-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-1 trials earlier.
n-2-back (post-deviation) | Baseline
  The n-2-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-2 trials earlier.
n-2-back (post-deviation) | 1 hour
  The n-2-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-2 trials earlier.
n-1-back (post-target) | Baseline
  The n-1-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-1 trials earlier.
n-1-back (post-target) | 1 hour
  The n-1-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-1 trials earlier.
n-2-back (post-target) | Baseline
  The n-2-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-2 trials earlier.
n-2-back (post-target) | 1 hour
  The n-2-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-2 trials earlier.
n-1-back (load) | Baseline
  The n-1-back (load) condition measures working memory performance under the cognitive demand of tracking stimuli 1 trial back.
n-1-back (load) | 1 hour
  The n-1-back (load) condition measures working memory performance under the cognitive demand of tracking stimuli 1 trial back.
n-2-back (post-load) | Baseline
  The n-2-back (post-load) condition assesses working memory performance on the trial immediately following a high cognitive load in the n-2-back task.
n-2-back (post-load) | 1 hour
  The n-2-back (post-load) condition assesses working memory performance on the trial immediately following a high cognitive load in the n-2-back task.
Coop-Wonka chart | Baseline
  The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Coop-Wonka chart | 1 hour
  The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 1 hour
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Pittsburgh Sleep Quality Index | Baseline
  The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 1 hour
  The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
State Trait Anxiety Inventory | Baseline
  The state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 1 hour
  The state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | Baseline
  The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 1 hour
  The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Epworth Sleepiness Scale | Baseline
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 1 hour
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Everyday Memory Errors Questionnaire | Baseline
  The Everyday Memory Errors Questionnaire is a brief self-report instrument designed to assess the frequency of memory lapses in daily life. It consists of multiple items that yield a total score reflecting the extent of everyday memory difficulties.
Everyday Memory Errors Questionnaire | 1 hour
  The Everyday Memory Errors Questionnaire is a brief self-report instrument designed to assess the frequency of memory lapses in daily life. It consists of multiple items that yield a total score reflecting the extent of everyday memory difficulties.
Falls Efficacy | Baseline
  The Falls Efficacy Scale is a brief self-report instrument designed to assess confidence in performing daily activities without falling. It consists of multiple items that yield a total score reflecting fear of falling and perceived fall-related self-efficacy.
Falls Efficacy | 1 hour
  The Falls Efficacy Scale is a brief self-report instrument designed to assess confidence in performing daily activities without falling. It consists of multiple items that yield a total score reflecting fear of falling and perceived fall-related self-efficacy.
Anterior-posterior balance | Baseline
  The maximum anterior-posterior displacement of the centre of pressure during a two-minute balance task.
Anterior-posterior balance | 1 hour
  The maximum anterior-posterior displacement of the centre of pressure during a two-minute balance task.
Medio-lateral balance | Baseline
  The maximum medio-lateral displacement of the centre of pressure during a two-minute balance task.
Medio-lateral balance | 1 hour
  The maximum medio-lateral displacement of the centre of pressure during a two-minute balance task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No